CLINICAL TRIAL: NCT02704585
Title: Comparison of Two Pulse Oximeters in Delivery Room: A Prospective Study
Brief Title: Comparison of Two Pulse Oximeters in Delivery Room
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Bromiker, Ruben M.D, Senior Neonatologist, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 118/15
Record Dates: First submitted 2016-02-24; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Hypoxia
Keywords: Neonatal resuscitation; Pulse oximetry
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nellcor (Other): Connection to Nellcor pulse oximeter for measuring oxygen saturation after birth
  Interventions: Device: Nellcor
- Masimo (Other): Connection to Masimo pulse oximeter for measuring oxygen saturation after birth
  Interventions: Device: Masimo

INTERVENTIONS:
Device: Nellcor — Measurement of pulse oximetry in the delivery room with Nellcor pulse oximeter
  Arms: Nellcor
Device: Masimo — Measurement of pulse oximetry in the delivery room with Masimo pulse oximeter
  Arms: Masimo

SUMMARY:
Time to stable reading of oxygen saturation at the delivery room will be compared between two different devices.

DETAILED DESCRIPTION:
After delivery babies will be located in the radiant warmer. The probe of each pulse oximeter will be applied to one of the feet. Both probes will be simultaneously connected to the female plug of the pulse oximeter.

Heart rate will be checked

Time to get a stable reading in each device (by observation on the devices' display) will be recorded; this will be the primary study outcome. Other vital signs (oxygen saturation, heart rate) and demographics) will be recorded as well.

Paired students T test will be used for the statistical analyzes.

ELIGIBILITY:
Inclusion Criteria:

* Neonates in the operation or delivery room immediately after delivery whose parents agreed to enter the study

Exclusion Criteria:

* Malformation of one of the legs, not allowing sensor application. Any situation in which the study might interfere with the treatment of the newborn

Ages: 1 Minute to 15 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Time to steady reading in the pulse oximeter | up to 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Bromiker, MD, Study Chair — Shaare Zedek Medical Center
Locations (1):
- Ruben Bromiker, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baquero H, Alviz R, Castillo A, Neira F, Sola A. Avoiding hyperoxemia during neonatal resuscitation: time to response of different SpO2 monitors. Acta Paediatr. 2011 Apr;100(4):515-8. doi: 10.1111/j.1651-2227.2010.02097.x. Epub 2011 Jan 17. PMID 21091987